CLINICAL TRIAL: NCT03025321
Title: Effects of Electrical Neuromodulation on Craving, Relapse and Cognitive Functions Among Patients With Cocaine Use Disorder: A Multi-Session tDCS Study
Brief Title: Effects of tDCS on Craving, Relapse and Cognitive Functions Among Patients With Cocaine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Ingmar Franken, Prof. Dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL57262.078.16
Record Dates: First submitted 2017-01-05; First posted 2017-01-19 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Cocaine Addiction
Keywords: Cocaine; tDCS; EMA; Inhibitory control; Reward processing; Addiction; dlPFC; craving; cognitive control
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transcranial direct current stimulation (Experimental): This group will receive bilateral tDCS (left cathodal/right anodal) over the DLPFC. The stimulation will take place two times daily for 13 minutes with a rest interval of 20 minutes for five consecutive days.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): The control group receives sham, for which the stimulator will be gradually turned off after 30 seconds.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — tDCS is an electrical brain stimulation method Participants will receive real-tDCS or sham twice daily for 13 min with an interval of 20 min for five consecutive days.

SUMMARY:
Repetitive bilateral (left cathodal/ right anodal) transcranial Direct Current Stimulation (tDCS) over the dorsolateral prefrontal cortex (DLPFC) reduces craving and seems to decrease relapse risk in addiction. However, little is known about the relapse rates in cocaine addiction after tDCS, despite the need for neurobiological treatments to reduce the high relapse rates in this population. The current study explores the effects of repetitive tDCS in a larger sample (N=60) of cocaine addicted patients on number of relapse days after three months. We expect that a decrease in relapse risk after tDCS is associated with cognitive control functioning. Therefore, risky decision making and inhibitory control will be measured before and after the interventions, and at three months follow-up. Ecological momentary assessment (EMA) will be used as a reliable measure for relapse, craving and mood.

DETAILED DESCRIPTION:
For this study, 60 cocaine addicted patients will receive real or sham bilateral tDCS (left cathodal/right anodal) over the DLPFC after one week in detox. The participants will receive this two times daily for 5 consecutive days. It is expected that this particular tDCS method will reduce relapse probability, as was previously seen in alcohol addicted patients. Furthermore, it is hypothesized that this therapeutic effect is associated with diminished craving and enhanced cognitive control. Craving, temptations and relapse, will be explored by means of Ecological Momentary Assessment (EMA). The mixed results in previous studies of tDCS on craving may be explained by the fact that craving in addiction is a momentary phenomenon which is difficult to reliably measure with more traditional methods like retrospective self-reports, for which EMA provides a solution. Cognitive control will be measured by means of inhibitory control during a Go/NoGo task and reward processing during a gambling task. The tasks will be performed at baseline, one day after the tDCS sessions and at three months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Meeting the DSM-V criteria for cocaine dependence
* The ability to speak, read, and write in Dutch at an eight-grade literacy level
* No severe withdrawal signs or symptoms at baseline

Exclusion Criteria:

* Indications of severe psychopathology (psychosis, severe mood disorder) as assessed by a physician
* A diagnosis of epilepsy, convulsions or delirium tremens during abstinence of cocaine use
* Any contraindication for electrical brain stimulation procedures such as electronic implants or metal implants
* Pregnancy or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Number of relapse days at three months follow-up | three months
  In an app on the smartphone participants can indicate when they relapsed at any time during 3 months starting from tDCS session 1. Participants will receive a reminder at the end of every week to fill this out.

SECONDARY OUTCOMES:
Number of relapse days at one week after the last tDCS session | 2 weeks
  In an app on the smartphone participants can indicate when they relapsed at any time during 2 weeks starting from tDCS session 1. Participants will receive a reminder at the end of every week to fill this out.
Craving | 2 weeks
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about craving for 2 weeks starting from tDCS session 1
Mood | 2 weeks
  Participants receive 4 prompts a day in the app on the smartphone to fill out questions about mood during 2 weeks starting from tDCS session 1
Inhibitory control | at baseline and one day after tDCS and at three months follow-up
  3 times measured by means of a cocaine related Go/NoGo task
Reward processing | at baseline and one day after tDCS and at three months follow-up
  3 times measured by means of a gambling task

CONTACTS AND LOCATIONS:
Locations (1):
- Antes, Rotterdam, Netherlands

REFERENCES:
- [Derived] Verveer I, van der Veen FM, Shahbabaie A, Remmerswaal D, Franken IHA. Multi-session electrical neuromodulation effects on craving, relapse and cognitive functions in cocaine use disorder: A randomized, sham-controlled tDCS study. Drug Alcohol Depend. 2020 Dec 1;217:108429. doi: 10.1016/j.drugalcdep.2020.108429. Epub 2020 Nov 23. PMID 33250383